CLINICAL TRIAL: NCT02146352
Title: AXIOS Stent With Electrocautery Enhanced Delivery System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xlumena, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP201303
Record Dates: First submitted 2014-05-13; First posted 2014-05-23 (Estimated); Results first posted 2015-10-02 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-09

CONDITIONS: Pancreatic Pseudocyst(s)
Keywords: Pancreatic pseudocyst
MeSH Terms: conditions — Pancreatic Pseudocyst

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): AXIOS Stent with Electrocautery Enhanced Delivery System
  Interventions: Device: AXIOS Stent with Electrocautery Enhanced Delivery System

INTERVENTIONS:
Device: AXIOS Stent with Electrocautery Enhanced Delivery System — Endoscopy with ultrasonography to implant AXIOS stent using electrocautery enhanced delivery system to allow drainage of pancreatic pseudocyst. Removal of AXIOS stent after 30 or 60 days.

SUMMARY:
The purpose of this study is to demonstrate the safety and effectiveness of the AXIOS Stent with Electrocautery Enhanced Delivery System for endoscopic transenteric drainage of pancreatic pseudocysts.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 75 years old, male or female
2. Eligible for endoscopic intervention
3. Acceptable candidate for endoscopic transluminal pancreatic pseudocyst drainage
4. Symptomatic pancreatic pseudocyst having the following characteristics:

   * Greater or equal to 6 cm in diameter (based upon the maximum cross-sectional area in the CT scan or transabdominal ultrasound).
   * Adherent to bowel wall, and
   * ≥70% fluid content
5. Patient understands the study requirements and the treatment procedures and provides written Informed Consent.
6. Patient is willing to comply with all specified follow-up evaluations, including willingness to undergo a pre/post CT imaging study.

Exclusion Criteria:

1. The fluid collection to be drained is an immature pseudocyst
2. The fluid collection to be drained is a cystic neoplasm
3. The fluid collection to be drained is a pseudoaneurysm
4. The fluid collection to be drained is a duplication cyst
5. The fluid collection to be drained is a non-inflammatory fluid collection
6. There is more than one pseudocyst requiring drainage
7. Abnormal coagulation:

   * INR > 1.5 and not correctable
   * presence of a bleeding disorder
   * platelets < 50,000/mm3
8. Altered anatomy that precludes the physician's ability to deliver the stent (decision on a case by case basis).
9. Intervening gastric varices or vessels within a one centimeter radius of the needle (visible using endoscopy or endoscopic ultrasound)
10. Any prior true anaphylactic reaction to contrast agents, nitinol (nickel titanium), silicone or any other materials contacting the patient.
11. Female of childbearing potential with a positive pregnancy test prior to the procedure or intends to become pregnant during the study.
12. Currently participating in another investigational drug of device study that has not completed the primary endpoint or that clinically interferes with the endpoints of this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-06; Primary Completion 2015-01 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven A Edmundowicz, MD, Principal Investigator — Washington University School of Medicine
Locations (8):
- United States (8):
  - University of Colorado Denver, Aurora, Colorado
  - Baptist Medical Center, Jacksonville, Florida
  - Florida Hospital, Orlando, Florida
  - Emory University, Atlanta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Washington University in St. Louis, St Louis, Missouri
  - Thomas Jefferson University, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment
Started | 30
30 or 60 Days Post-procedure | 30
7 Days Post-stent Removal | 28
Completed | 28
Not Completed | 2
Not completed — Death | 1
Not completed — Patient entered hospice care | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.0 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 17
Region of Enrollment [Number; unit: participants]
  United States | 30
Height [Mean (Standard Deviation); unit: inches] | 67.3 (4.3)
Weight [Mean (Standard Deviation); unit: pounds] | 172.9 (36.8)

OUTCOME MEASURES:

1. Primary Outcome: Safety/Adverse Event Outcome Measure 1
Description: Freedom from access site-related bleeding requiring transfusion
Time Frame: Index procedure through 1-week post-stent removal
Population: Entire patient cohort
Measure: Number; unit: percentage of patients
Arm/Group | Treatment
Number analyzed (Participants) | 30
percentage of patients | 100

2. Secondary Outcome: Stent Retention Outcome Measure
Description: Stent Retention: The stent must remain in place for up to 60 days
Time Frame: 30 or 60 days post-procedure
Population: Per Protocol Population
Measure: Number; unit: percentage of patients
Arm/Group | Treatment
Number analyzed (Participants) | 30
percentage of patients | 100

3. Secondary Outcome: Lumen Patency Outcome Measure
Description: Lumen Patency: The stent lumen must be patent at 30 days and/or 60 days of implantation.
Time Frame: 30 and/or 60 days post-procedure
Population: Per Protocol
Measure: Number; unit: percentage of patients
Arm/Group | Treatment
Number analyzed (Participants) | 30
percentage of patients | 86.7

4. Secondary Outcome: Technical Success Outcome Measure 1
Description: Technical success: Successful placement of the AXIOS stent using the Electrocautery Enhanced AXIOS Delivery System
Time Frame: Index Procedure
Population: Per Protocol
Measure: Number; unit: percentage of patients
Arm/Group | Treatment
Number analyzed (Participants) | 30
percentage of patients | 100

5. Secondary Outcome: Clinical Success Outcome Measure
Description: Clinical success: At least a 50% decrease in pseudocyst size at 30 days or 60 days
Time Frame: 30 or 60 days post-procedure
Population: Entire patient cohort
Measure: Number; unit: percentage of patients
Arm/Group | Treatment
Number analyzed (Participants) | 30
percentage of patients | 83.3

6. Primary Outcome: Safety/Adverse Event Outcome Measure 2
Description: Freedom from access site-related infection requiring intravenous or intramuscular antibiotics and/or extended hospitalization
Time Frame: Index procedure through 1-week post-stent removal
Population: Entire patient cohort
Measure: Number; unit: percentage of patients
Arm/Group | Treatment
Number analyzed (Participants) | 30
percentage of patients | 100

7. Primary Outcome: Safety/Adverse Event Outcome Measure 3
Description: Freedom from surgery for access-site related perforation
Time Frame: Index procedure through 1-week post-stent removal
Population: Entire patient cohort
Measure: Number; unit: percentage of patients
Arm/Group | Treatment
Number analyzed (Participants) | 30
percentage of patients | 100

8. Primary Outcome: Safety/Adverse Event Outcome 4
Description: Freedom from stent migration/dislodgement into the pseudocyst or enteral lumen
Time Frame: Index procedure through 1-week post-stent removal
Population: Patients for which AXIOS stent migration/dislodgement could be assessed
Measure: Number; unit: percentage of patients
Arm/Group | Treatment
Number analyzed (Participants) | 28
percentage of patients | 96.4

9. Primary Outcome: Safety/Adverse Event Outcome Measure 5
Description: Freedom from tissue injury, defined as ulceration at site of stent implant as observed to persist through 1-week post-stent removal
Time Frame: Index procedure through 1-week post-stent removal
Population: Patients for which AXIOS stent was removed and tissue at site of stent implant was observed at time of removal
Measure: Number; unit: percentage of patients
Arm/Group | Treatment
Number analyzed (Participants) | 28
percentage of patients | 100

10. Primary Outcome: Safety/Adverse Event Outcome Measure 6
Description: Freedom from serious adverse event associated with the AXIOS stent and/or (index) implant procedure
Time Frame: Index procedure through 1-week post-stent removal
Population: Entire patient cohort
Measure: Number; unit: percentage of patients
Arm/Group | Treatment
Number analyzed (Participants) | 30
percentage of patients | 93.3

11. Secondary Outcome: Technical Success Outcome Measure 2
Description: Technical Success: Successful removal of AXIOS stent using standard endoscopic snare or forceps
Time Frame: 30 or 60 Day Post-procedure
Population: Per Protocol
Measure: Number; unit: percentage of patients
Arm/Group | Treatment
Number analyzed (Participants) | 27
percentage of patients | 100

ADVERSE EVENTS:
Time Frame: Index procedure through 1-week post-stent removal
Arm/Group | Treatment
Serious Adverse Events (participants affected / at risk) | 13/30
Other Adverse Events (participants affected / at risk) | 10/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=30)
Pancreatitis (Gastrointestinal disorders) | 9 (10)
Bronchitis (Infections and infestations) | 1 (1)
Biliary Stricture (Hepatobiliary disorders) | 1 (1)
Bleeding post-AXIOS stent removal (Surgical and medical procedures) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (2)
Chest pain/shortness of breath (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=30)
Abdominal Pain (Gastrointestinal disorders) | 3 (3)
Ascites (Gastrointestinal disorders) | 1 (1)
Bleeding post-AXIOS stent removal (Surgical and medical procedures) | 1 (1)
Blood in urine (Renal and urinary disorders) | 1 (1)
Chest pain (Cardiac disorders) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1)
Fever (Infections and infestations) | 1 (1)
Lightheadedness/ dizziness (General disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Pancreatic duct leak (Endocrine disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Spontaneous stent migration (Gastrointestinal disorders) | 1 (1)
Ulceration (Gastrointestinal disorders) | 1 (1)
Weight loss (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI must wait 9 months after close of study for Sponsor to present collaborative publication. If Sponsor does not publish within 9 months after close of study, PI may publish institution's results at that time. Sponsor can review results prior to public release and embargo communications on trial results for a period that is more than 60 days but less than or equal to 6 months from the date the PI gets the objection. The Sponsor cannot require changes to the communication nor extend the embargo.